CLINICAL TRIAL: NCT02014961
Title: Worm Study: Identification of Modifier Genes in a Unique Founder Population With Sudden Cardiac Death
Brief Title: Worm Study: Modifier Genes in Sudden Cardiac Death
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: METC 142060
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Brugada Syndrome; Long QT Syndrome 3
MeSH Terms: conditions — Brugada Syndrome; Long Qt Syndrome 3 | interventions — Exome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mutation Carriers (Active Comparator): Whole-exome sequencing (WES) Dermal biopsy Gastro-intestinal questionnaire
  Interventions: Procedure: Dermal biopsy; Behavioral: Gastro-intestinal questionnaire; Genetic: Whole-exome sequencing
- Non-Mutation Carriers (Placebo Comparator): Whole-exome sequencing (WES) Gastro-intestinal questionnaire
  Interventions: Behavioral: Gastro-intestinal questionnaire; Genetic: Whole-exome sequencing
- Spouse (Other): Whole-exome sequencing (WES) 12-Lead ECG
  Interventions: Genetic: Whole-exome sequencing

INTERVENTIONS:
Procedure: Dermal biopsy — Skin biopsy
  Arms: Mutation Carriers
Behavioral: Gastro-intestinal questionnaire — Pagi-Sym, Bristol Stool Chart, gastrointestinal symptom rating scale (GSRS)
  Arms: Mutation Carriers; Non-Mutation Carriers
Genetic: Whole-exome sequencing — Whole-exome sequencing (WES)

SUMMARY:
Quest for modifier genes associated with ventricular arrhythmias in presence of a cardiac sodium channel gene (SCN5A-delPhe1617) mutation.

DETAILED DESCRIPTION:
In a large Dutch SCN5A founder population with malignant ventricular arrhythmias, the investigators aim to identify genetic modifiers by means of whole-exome sequencing and to establish a comprehensive genotype-phenotype correlation, focussing on clinical and cellular electrophysiological characteristics and neurocardiac modulation.

ELIGIBILITY:
Inclusion Criteria (mutation carrier group):

* Age ≥ 18 years.
* Heterozygous or homozygous carriership of SCN5A-delPhe1617.
* Confirmed kinship to the founder population by haplotype analysis using predefined microsatellite markers.
* Written informed consent.

Inclusion Criteria (non-mutation carrier group):

* Age ≥ 18 years.
* Non SCN5A-delPhe1617 genotype.
* Confirmed kinship to the Founder Group by haplotype analysis using predefined microsatellite marker.
* Written informed consent.

Inclusion criteria Spouse Group

* Age ≥ 18 years.
* Biological parent of SCN5A-delPhe1617 positive subject participating to the Worm Study, and not belonging to study group 1 or 2.
* Written informed consent.

Exclusion Criteria:

* Age ≥ 18 years.
* Biological parent of SCN5A-delPhe1617 positive subject participating to the Worm Study, and not belonging to study group 1 or 2.
* Written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Estimated)
Dates: Start 2015-04; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Difference in genetic profile (e.g. modifier genes) between mutation carriers expressing different phenotypes and non-mutation carriers. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Volders, M.D., Ph.D., Study Director — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands